CLINICAL TRIAL: NCT02350920
Title: A Randomized Controlled Trial of Acceptance and Commitment Therapy (ACT) in Inflammatory Bowel Disease
Brief Title: Acceptance and Commitment Therapy (ACT) in Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Hugh Mulcahy, Professor Hugh Mulcahy, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UCDublin
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; Crohn's disease; ulcerative colitis; ACT
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Committment Therapy (ACT) (Active Comparator): This group will consist of patients who will receive ACT therapy.This intervention will run with 8-12 participants in each group for a duration of 8 weeks. Each group session will last 1-1.5 hours.
  Interventions: Behavioral: Acceptance and Committment Therapy (ACT)
- Control (No Intervention): The control group will consist of patients who will receive no ACT therapy during the 26 week st udy period

INTERVENTIONS:
Behavioral: Acceptance and Committment Therapy (ACT) — This intervention will run with 12-15 participants in each group for a duration of 8 weeks. Each group session will last 1-1.5 hours.
  Other Names: ACT
  Arms: Acceptance and Committment Therapy (ACT)

SUMMARY:
Over 18,000 Irish people are affected by the inflammatory bowel diseases (IBD), Crohn's disease and ulcerative colitis. These illnesses often arise at a young age and can be associated with significant physical disability. In addition, there is considerable psychosocial disability associated with IBD. Previous studies have suggested that simple psychological interventions may be valuable in improving quality of life and may even improve disease activity. However, there has been no comprehensive trial to determine the precise effect of psychological interventions on quality of life (QOL), stress or disease activity. Our aim is to conduct a randomised controlled trial of a simple psychological intervention to determine it's effect on QOL and stress

DETAILED DESCRIPTION:
The inflammatory bowel diseases (IBD), which include Crohn's disease and ulcerative colitis, are chronic conditions that often arise in young patients and may lead to a lifetime of physical disability. Psychological disabilities are also prevalent in patients with chronic diseases and epidemiological studies indicate that IBD patients are at increased risk of anxiety and mood disorders, with depression rates more than double that of matched community samples (27% versus 12%). IBD patients are also at increased risk of illness-related psychological difficulties including body image concerns, sexual problems and reduced self-esteem.

Therapeutic approaches to inflammatory bowel disease naturally focus on treatments that minimise disease activity and normalise physical function. Thus, there has been considerable research conducted on 5 ASA medications, steroids, immune modulators and biologic agents. In contrast, little attention has been paid to important, but 'low-technology', issues including quality of life and psychological comorbidities including depression, anxiety, stress, altered body image, sexuality, illness attitudes, self-esteem and other psychosocial IBD co-morbidities. Nevertheless, patient reported data and outcomes are increasingly being incorporated into research that informs strategic healthcare documents that, in turn, help formulate healthcare policy. Contemporary European and British guidelines now emphasise the benefits of a patient centred service that supplies psychological as well as medical support.

In addition to the burden that psychological disease places upon IBD patients, there is evidence that psychological morbidity and stress is also associated with disease activity. IBD patients with depression experience more disease flares than those with no diagnosable psychological condition and a Canadian study has also suggested that stress can be associated with disease flares. In contrast, a Spanish study on 163 patients concluded that stressful life events do not trigger exacerbations in IBD patients. Overall, it is likely that the relationship between stress and disease activity is bi-directional with each one influencing the other to some extent.

To date, interventions aimed at reducing psychological distress in IBD have tended to focus on either psychological education, stress management including relaxation techniques and autogenic training, psychodynamic psychotherapy, cognitive behavioral therapy and hypnosis. Studies have been variable with regard to psychological content and almost all had multiple methodological limitations, making it difficult to draw conclusions about the value of these interventions. Perhaps the most comprehensive review of psychological studies in IBD, which included 16 studies, concluded that while psychological interventions can make a positive contribution to best practice multidisciplinary IBD treatment, well designed studies are needed to determine the efficacy of different treatments.

We aim to conduct a multicenter randomised controlled trial to determine the efficacy of Acceptance and Commitment Therapy (ACT) on the psychological wellbeing of IBD patients.

We aim to include 80 patients in this longitudinal study (40 in each arm). IBD patients attending St Vincent's University Hospital and Beaumont Hospital are treated in protocol driven inflammatory bowel disease clinics with therapy adhering to international treatment guidelines. We currently use protocols developed by the European Crohn's and Colitis Organisation (ECCO) and American Gastroenterology Association (AGA). Our care incorporates formalised multidisciplinary teamwork with standardised clinical monitoring, use of contemporary biomarkers of disease activity and a full range of current therapies including 5-ASA and steroid medications, immunological therapies, open and laparoscopic surgery as appropriate, endoscopic treatment as necessary and the latest biological agents as per protocol. Thus, the study will take place in a clinical environment in which we adhere to the most modern practices.

Initial assessment

1. Biological assessment

   The initial assessment will comprise standardised and validated questionnaires to determine biological status. Specifically, we will assess:

   Demographic data Region, urban/rural, race, age, education, martial status, family history, occupation, employment status, smoking and alcohol history Nutritional status Body Mass Index Exercise status Godin Leisure-Time Exercise Questionnaire IBD history Disease type, duration, clinical, therapeutic and surgical history, Hospital admissions and visits, GP visits Disease activity Harvey Bradshaw Index (CD), Mayo Score (UC), physical examination Medication adherence Medication Adherence Report Scale 5 (MARS5) Laboratory indices Biochemical, immunological and haematological variables, faecal calprotectin, hair cortisol
2. Psychological assessment

This will include validated instruments to build a structured picture of the IBD illness. We will assess:

General Quality of Life Short Form 12, Healthy days IBD specific QOL Short Health Scale Stress/anxiety/depression Depression Anxiety Stress Scales (DASS) 21 and Stress Thermometer Self Esteem Rosenberg Self Esteem Survey Body Image Modified Hopwood Body Image Scale Disease acceptance Acceptance and Action Questionnaire - Revised

Interventions Group 1) Control (n=40) The control group will consist of 40 patients who will who will not receive treatment for 26 weeks and will then receive the ACT program.

Group 2) Acceptance and Commitment therapy (n=40) ACT is a behavioural therapeutic approach that uses processes of acceptance, mindfulness, commitment and behaviour change to increase psychological flexibility. In terms of ACT for IBS specifically, its use is in guiding patients to develop a willingness to come in contact with their unpleasant experiences of physical symptoms and with the feeling of embarrassment, anticipatory anxiety and distressing thoughts commonly associated with IBS. The former agenda of trying to eliminate symptoms and distressing cognitive and emotional states can then be replaced by an agenda focusing on creating a more meaningful life with IBS.

Assessments during intervention period Weekly assessments will be performed during the intervention period. These will include the Harvey Bradshaw Index (CD), Mayo Score (UC), Short Health Scale, (DASS) 21 and Stress Thermometer

Eight week assessment

1. Biological assessment Medication adherence Medication Adherence Report Scale 5 (MARS5) Nutritional status Body Mass Index Exercise status Godin Leisure-Time Exercise Questionnaire Disease activity indices Harvey Bradshaw Index (CD), Mayo Score (UC) Laboratory indices Biochemical, immunological and haematological variables, faecal calprotectin, hair cortisol
2. Psychological assessment General Quality of Life Short Form 12, Healthy days IBD specific QOL Short Health Scale Anxiety/Depression Beck Depression Inventory, Beck Anxiety Inventory Stress Depression Anxiety Stress Scales (DASS) 21 and Stress Thermometer Self Esteem Rosenberg Self Esteem Survey Body Image Modified Hopwood Body Image Scale Sexuality Modified Golombok-Rust Inventory Disease acceptance Acceptance and Action Questionnaire - Revised

26 week assessment Repeat of 8 week assessment

Hair Cortisol Measurement The effects of stress are mediated by the stress hormone cortisol. Cortisol is involved in the regulation of glucose and lipid metabolism, body composition, and the immune system. Cortisol is traditionally measured in serum or saliva. However, because cortisol is secreted in a circadian rhythm and with pulses, the timing of sample collection is crucial when measuring cortisol in serum or saliva. In addition, cortisol is a stress hormone, and acute stress, such as that caused by the research setting or venepuncture, will influence measurements. A single measurement of cortisol in serum or saliva therefore poorly reflects medium and long-term cortisol levels. An alternative method to measure cortisol is in scalp hair. This method offers long-term measurements of cortisol levels, with 1cm of hair representing cortisol levels of approximately one month. In the last few years, the measurement of cortisol in scalp hair has been well validated. We will measure hair cortisol at the initial assessment, at the conclusion of therapy (8 weeks) and at the 26 week visit.

ELIGIBILITY:
Inclusion Criteria:

* IBD patients who have inactive disease and either a stressometer score of ≥5 or a Short Health Scale score of ≥80 will be eligible for inclusion

Exclusion Criteria:

* Patients under 18 years,
* Patients over 65 years,
* pregnant females,
* patients currently attending psychiatric services,
* patients currently receiving antidepressant medication,
* patients who have received steroid medications in the past three months,
* patients who have previously undergone a stress management programme (relaxation techniques, autogenic training, psychodynamic psychotherapy, cognitive behavioural therapy, hypnosis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Changes in stress measured by the Depression, Anxiety and Stress Scale (DASS 21) | 20 weeks
  Changes in stress measured by the Depression, Anxiety and Stress Scale (DASS 21)

SECONDARY OUTCOMES:
Changes in quality of life measured by the Short Health Scale (SHS) | 20 weeks
  Changes in quality of life measured by the Short Health Scale (SHS)
Changes in disease activity measured by the Short Mayo Scale and Harvey Bradshaw Index | 20 weeks
  Changes in disease activity measured by the Short Mayo Scale and Harvey Bradshaw Index
Changes in hair cortisol levels | 20 weeks
  Changes in hair cortisol levels
Changes in medication requirements | 20 weeks
  Changes in need for medications including steroids, immunomodulators and biologic agents over the study period
Changes in General and GUT specific inflammatory markers | 20 weeks
  Changes in CRP and faecal calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: hugh mulcahy, md, Principal Investigator — UCD
Locations (1):
- St Vincent's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available for other researchers following publication of of our results in the medical literature. A datafile may be obtained by contacting Prof. Hugh Mulcahy at hemulc@hotmail.com, giving details of i) proposed use of the data and ii) what form of acknowledgement of the data will be made by the researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available one month following publication, estimated to be February 2019 and will be made available for a period of five years
Access Criteria: IPD will be available as an excel file to researchers on application to Professor Hugh Mulcahy at hemulc@hotmail.com, specifying the nature of the analyses to be performed with these data and details of acknowledgements to be made regarding the data. No type of analysis will be excluded from consideration

REFERENCES:
- [Background] Elkjaer M, Moser G, Reinisch W, Durovicova D, Lukas M, Vucelic B, Wewer V, Frederic Colombel J, Shuhaibar M, O'Morain C, Politi P, Odes S, Bernklev T, Oresland T, Nikulina I, Belousova E, Van der Eijk I, Munkholm P. IBD patients need in health quality of care ECCO consensus. J Crohns Colitis. 2008 Jun;2(2):181-8. doi: 10.1016/j.crohns.2008.02.001. Epub 2008 Apr 9. PMID 21172209
- [Background] Mittermaier C, Dejaco C, Waldhoer T, Oefferlbauer-Ernst A, Miehsler W, Beier M, Tillinger W, Gangl A, Moser G. Impact of depressive mood on relapse in patients with inflammatory bowel disease: a prospective 18-month follow-up study. Psychosom Med. 2004 Jan-Feb;66(1):79-84. doi: 10.1097/01.psy.0000106907.24881.f2. PMID 14747641
- [Background] Bitton A, Sewitch MJ, Peppercorn MA, deB Edwardes MD, Shah S, Ransil B, Locke SE. Psychosocial determinants of relapse in ulcerative colitis: a longitudinal study. Am J Gastroenterol. 2003 Oct;98(10):2203-8. doi: 10.1111/j.1572-0241.2003.07717.x. PMID 14572569
- [Background] Vidal A, Gomez-Gil E, Sans M, Portella MJ, Salamero M, Pique JM, Panes J. Life events and inflammatory bowel disease relapse: a prospective study of patients enrolled in remission. Am J Gastroenterol. 2006 Apr;101(4):775-81. doi: 10.1111/j.1572-0241.2006.00476.x. Epub 2006 Feb 22. PMID 16494590
- [Background] Knowles SR, Monshat K, Castle DJ. The efficacy and methodological challenges of psychotherapy for adults with inflammatory bowel disease: a review. Inflamm Bowel Dis. 2013 Nov;19(12):2704-15. doi: 10.1097/MIB.0b013e318296ae5a. PMID 23846488
- [Background] Gow R, Thomson S, Rieder M, Van Uum S, Koren G. An assessment of cortisol analysis in hair and its clinical applications. Forensic Sci Int. 2010 Mar 20;196(1-3):32-7. doi: 10.1016/j.forsciint.2009.12.040. Epub 2010 Jan 21. PMID 20096513
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Wynne B, McHugh L, Gao W, Keegan D, Byrne K, Rowan C, Hartery K, Kirschbaum C, Doherty G, Cullen G, Dooley B, Mulcahy HE. Acceptance and Commitment Therapy Reduces Psychological Stress in Patients With Inflammatory Bowel Diseases. Gastroenterology. 2019 Mar;156(4):935-945.e1. doi: 10.1053/j.gastro.2018.11.030. Epub 2018 Nov 16. PMID 30452919